CLINICAL TRIAL: NCT01502163
Title: Efficacy of a Convective Prewarming System in Prevention of Perioperative Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Collaborators: UZ Gent, Belgium (Unknown); Policlinica de Guipuzcoa, San Sebastian, Spain (Unknown)
Responsible Party: Principal Investigator, Dr. T. Perl, Principal investigator, University of Göttingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/4/11
Record Dates: First submitted 2011-12-23; First posted 2011-12-30 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Perioperative Hypothermia
Keywords: perioperative hypothermia; prewarming; forced air warming; insulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): * No prewarming
  * Intraoperative forced air warming (Thermoflect™/Mistral Air™) (after induction of anaesthesia, before surgery starting)
  * Passive insulation with Thermoflect™ material.
  * All fluids administrated intraoperative will be warmed.
- Group passive prewarming (Active Comparator): * Passive prewarming / insulation on nursery ward before transport to the OR (Thermoflect TSCI, Amersfoort, NL)
  * Intraoperative forced air warming (Thermoflect™ / Mistral Air ™) The forced air warming will be applied after induction of anaesthesia.
  * All fluids administrated intraoperative will be warmed.
  Interventions: Device: Thermoflect [TM] passive insulation
- Group Active prewarming (Active Comparator): * Active prewarming on nursery ward before transport to the OR (Thermoflect™/Mistral Air™, TSCI, Amersfoort, NL)
  * Intraoperative forced air warming (Thermoflect™ / Mistral Air ™) The forced air warming will be applied after induction of anaesthesia.
  * All fluids administrated intraoperative will be warmed.
  Interventions: Device: Active prewarming (Thermoflect™/Mistral Air™, TSCI, Amersfoort, NL)

INTERVENTIONS:
Device: Thermoflect [TM] passive insulation — passive insulation in the preoperative phase, befor induction of anesthesia
  Arms: Group passive prewarming
Device: Active prewarming (Thermoflect™/Mistral Air™, TSCI, Amersfoort, NL) — Prewarming Thermoflect™/Mistral Air™, TSCI, Amersfoort, NL before induction of anesthesia
  Arms: Group Active prewarming

SUMMARY:
Although several measures for prevention of perioperative hypothermia have been introduced the last decades, perioperative hypothermia is still a frequent complication and associated with a negative outcome.

For not long lasting surgery without specific risk for hypothermia the standard procedure for prevention of perioperative hypothermia is insulation. However, the insulation is often not effective enough to prevent intra- and postoperative hypothermia. The implementation of a prewarming is difficult because of variable OR schedules and therefore not often applied.

In the planed prospective, multicenter, randomised-controlled trial will the efficacy of a convective prewarming system on prevention of intra- and perioperative hypothermia (Thermoflect™, TSCI, Amersfoort, NL) be compared to an intraoperative application of forced air warming with or without passive insulation before induction of anesthesia.

The studied prewarming device is easy to use and will be applied on the nursery ward 30-60 minutes before transfer of the patient to the OR.

Perioperative hypothermia is a common complication in general aesthesia. Perioperative hypothermia is associated with medical risks as intraoperative impaired coagulation due to reversible platelet dysfunction, a prolonged bleeding time and increased intraoperative blood loss. In the postoperative course the perioperative hypothermia is especially for patients with cardiopulmonary diseases a relevant problem. Not at least sensual cold and shivering is uncomfortable for the patient.

The study is conducted as a multicenter, prospective, randomised controlled trial. All patients will receive intraoperatively a forced air warming device (Termoflect™/Mistral Air ™). For one intervention group will additionally the insulation with the Thermoflect™ will be applied on nursery ward, the second intervention group will receive additionally a convective air warmer/ reflective blanket (Thermoflect™/Mistral Air™, TSCI, Amersfoort, NL) preoperatively on study day on nursery ward.

The aim of the study is to prove the hypothesis that a preoperative insulation with a commercial insulation material (Thermoflect™, TSCI, Amersfoort, NL) leads to a lower incidence of perioperative hypothermia in general anesthesia. The second hypothesis is, that an active prewarming (Thermoflect™ with Mistral Air™, TSCI, Amersfoort, NL) is associated with a more less incidence of periopative hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 75 years
* BMI from 20 to 30 kg/m2
* Risk class ASA I to III
* Scheduled time for surgery 30 to 120 minutes
* Scheduled anaesthesia with remifentanil, propofol, rocuronium and sevofluran
* Ability of informed consent

Exclusion Criteria:

* Adipositas permagna
* Risk class ASA IV to V
* Hypo- and Hyperthyroidism
* Febrile infection
* Pregnancy
* Scheduled time for surgery < 30 or > 120 minutes
* Known incompatibility for midazolam, remifentanil, propofol oder rocuronium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Core Temperature at end of surgery | Approximatly 120 minutes (at end of surgery)

SECONDARY OUTCOMES:
Number of patients with intraoperative hypothermia (Core temperature < 36°C). | Approximatly 120 minutes (at end of surgery)
Oral temperature before induction of anaesthesia | at induction of anesthesia
Temperature at arrival in the recovery room | Approximatly 140 minutes after induction (at arrival in recovery room)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Quintel, Prof, Study Chair — University Göttingen, Germany; Thorsten Perl, MD, Principal Investigator — University Göttingen, Germany; Koen Reyntjens, MD, Principal Investigator — UZ Gent, Belgium; Juan Zamballos, Prof., Principal Investigator — Policlinica de Guipuzcoa, San Sebastian, Spain
Locations (3):
- UZ Gent, Ghent, Belgium
- Department of Anesthesiology, Emergency- and Intensive Care Medicine, Göttingen, Germany
- Policlinica de Guipuzcoa, Donostia / San Sebastian, Spain